CLINICAL TRIAL: NCT00991861
Title: Double-blind, Randomized, Multi-centre Phase II Study to Evaluate the Efficacy and Safety of Topically Applied LAS41007 Once Daily and LAS41007 Twice Daily Versus LAS106521 Gel Twice Daily in the Treatment of Actinic Keratosis Grade I to II
Brief Title: Efficacy and Safety Study of LAS41007 in the Treatment of Actinic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H 569 000 - 0908; EudraCT: 2009-012063-33
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; AK; NMSC
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LAS41007 o.d. (Experimental): Once daily
  Interventions: Drug: LAS41007 o.d.
- LAS41007 b.i.d. (Experimental): Twice daily
  Interventions: Drug: LAS41007 b.i.d.
- LAS106521 (Active Comparator)
  Interventions: Drug: LAS106521

INTERVENTIONS:
Drug: LAS41007 o.d. — Once daily, topical application
  Arms: LAS41007 o.d.
Drug: LAS41007 b.i.d. — Twice daily, topical application
  Arms: LAS41007 b.i.d.
Drug: LAS106521 — Twice daily, topical application
  Arms: LAS106521

SUMMARY:
The aim of this study is to determine the efficacy, safety and tolerability of either a once or twice daily topical application of LAS41007 compared to a twice daily application of LAS106521 in the treatment of actinic keratosis.

ELIGIBILITY:
Inclusion Criteria:

* At least 4-10 clinically assessed actinic keratosis grade I to II (according to Olsen et al, 1991) in the face/forehead and/or on the bald scalp
* The diameter of each AK target lesion is not less than 0.5 cm and not greater than 1.5 cm
* The target lesions must be located in overall 2 treatment areas with a size of 25 cm2 per treatment area

Exclusion Criteria:

* Have evidence of clinically significant or unstable medical conditions such as:

  * metastatic tumor or tumor with high probability of metastatic spread
  * heart failure (NYHA class III or higher)
  * immunosuppressive disorder (e.g. HIV)
  * hematologic, hepatic, renal, neurologic or endocrine disorder.
  * collagen-vascular disorder (e.g. cerebrovascular disorder or other bleedings).
  * gastrointestinal disorder (e.g. active ulcera or history of recurrent peptic ulcera or hemorrhage)
* Suffer from paresthesia in the treatment areas
* Show Cornu cutaneum of the skin and/or hypertrophic AK lesions in the treatment areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Histological clearance of one pre-selected target lesion | Day 120
Complete clinical clearance of all target lesions in the treatment areas | Day 120

SECONDARY OUTCOMES:
Physician's Global Tolerability Assessment (PGT) | Day 120

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Willers, MD, MBA, Study Director — Almirall Hermal GmbH
Locations (1):
- Investigational Site, Hamburg, Germany

REFERENCES:
- See also: Almirall Corporate Website — http://www.almirall.com/webcorp2/cda/ImD_04_02.jsp